CLINICAL TRIAL: NCT03202186
Title: Double-Blind Trial Investigating the Efficacy of Different Doses of Progesterone Compared With Placebo for Treatment of Vasomotor Symptoms
Brief Title: Study of Progesterone in Treatment of Vasomotor Symptoms
Acronym: PROGEST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to recruit subjects
Sponsor: BHR Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHR-401-301
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Menopause Related Conditions
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Placebo controlled parallel arm study for 12 weeks
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): oral administration of Placebo capsule
  Interventions: Drug: Placebo oral capsule
- Progesterone 200 mg (Experimental): oral administration of progesterone 200 mg
  Interventions: Drug: Progesterone oral capsule
- Progesterone 300 mg (Experimental): oral administration of progesterone 300 mg
  Interventions: Drug: Progesterone oral capsule
- Progesterone 400 mg (Experimental): oral administration of progesterone 400 mg
  Interventions: Drug: Progesterone oral capsule

INTERVENTIONS:
Drug: Progesterone oral capsule — Oral capsule treatment
  Arms: Progesterone 200 mg; Progesterone 300 mg; Progesterone 400 mg
Drug: Placebo oral capsule — Oral capsule treatment
  Arms: Placebo

SUMMARY:
The primary objective of the clinical trial is to demonstrate superiority of BHR401 (oral micronized progesterone) versus placebo as a monotherapy for moderate to severe VMS in postmenopausal women. Three different doses of BHR-401 (200 mg, 300 mg or 400 mg) will be tested against placebo in hierarchical order, starting with the highest dose. Superiority will be defined as a significant (significance level α = 0.05) reduction of moderate to severe VMS frequency compared to placebo at treatment week 12 (the primary efficacy endpoint of the study).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Adult (≥ 18 years), postmenopausal women, where postmenopause is defined as

  * at least 12 months of spontaneous amenorrhea, or
  * 6 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) levels > 40 mIU/ml, or
  * status at least 6 weeks after bilateral oophorectomy with or without hysterectomy
* Non-smoker
* Mammography without pathological findings obtained within routine medical care no longer than 12 months prior to screening visit
* Cervical smear (Papanicolaou test) without pathological findings (i.e. < III) obtained no longer than 12 months prior to screening visit
* In addition subjects need to fulfil the following criterion in order to be randomized (i.e. to enter the treatment period):

  * A minimum of 50 moderate to severe VMS episodes over the last 7 consecutive days prior to the baseline visit, as documented in the patient diary.

Exclusion Criteria:

* Use of any hormone replacement therapy (including phytoestrogens and other plant-derived sex hormones) during the previous 12 weeks prior to screening
* Ongoing or suspicion of any estrogen-dependent malignancy.
* Endometrial thickness ≥ 5 mm at screening visit
* Any history or current presence or suspicion of breast cancer, including carcinoma in situ and other pre-cancerous conditions
* Active malignant disease of any organ system (except for basal localized basal cell carcinoma of the skin) or history thereof in the last 5 years prior to screening visit
* Vaginal bleeding due to unidentified reason within 6 weeks prior to screening
* Ongoing venous thromboembolic event or history thereof within 12 months prior to screening visit
* Known severe renal insufficiency (defined as glomerular filtration rate, GFR < 30 mg/min/1.73 m²) at screening visit
* Known lipid metabolism disturbances of genetic origin (e.g. familial hypercholesterolemia, familial hypertriglyceridemia)
* Acute or chronic liver diseases or a history of liver disease with liver enzymes having not normalized since then
* Severe disturbances of hepatic function (including porphyria), hepatic tumors, also in medical history
* Rotor syndrome or Dubin-Johnson syndrome
* History of icterus or generalized pruritus during a previous pregnancy
* History of myocardial infarction, stroke or transient ischemic attack or severe cardiac disease, including symptomatic chronic heart failure
* Ongoing major depression
* Subjects who currently take or are planned to commence treatment with SSRI, SNRI for any reason during the course of the study
* Diabetes mellitus
* Hypersensitivity to progesterone or excipients (e.g. soy) of the study medication
* Medical history of HIV infection
* Concomitant diseases or therapies that may cause VMS or affect VMS frequency or severity, e.g. but not limited to poorly controlled thyroid dysfunction (thyroid medication should be stable for at least 12 weeks prior to screening and TSH levels should be within range), fear disorders (e.g. panic disorders)
* Participation in a clinical trial or intake of any investigational medicinal product within three months prior to screening visit
* Previous participation in this clinical trial
* Known or suspected drug or alcohol abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Frequency of moderate to severe vasomotor symptoms at 12 weeks | 12 weeks
  the change vs. baseline of the frequency of moderate or severe VMS episodes (per day) after 12 weeks of treatment with BHR-401or placebo

SECONDARY OUTCOMES:
Frequency of moderate to severe vasomotor symptoms at 4 weeks | 4 weeks
  the change vs. baseline of the frequency of moderate or severe VMS episodes (per day)
Severity of vasomotor symptoms at 12 weeks | 12 weeks
  the change vs. baseline of the secerity of moderate or severe VMS episodes (per day)
Severity of vasomotor symptoms at 4 weeks | 4 weeks
  the change vs. baseline of the severity of moderate or severe VMS episodes (per day)

OTHER OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 12 weeks
Kupperman Index | 4 and 12 weeks
  Change vs. baseline of postmenopausal symptoms as assessed by the physician by means of the Kupperman Index inventory after 4 weeks and 12 weeks of treatment
Sleep quality assessed by means of the Pittsburgh Sleep Quality Index (PSQI) | 4 and 12 weeks
  Change in subjective sleep quality vs. baseline as assessed by means of the Pittsburgh Sleep Quality Index (PSQI) after 4 weeks and 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development, PhD, Study Director — BESINS Healthcare Ireland Ltd.
Locations (1):
- Fachärztin für Gynäkologie und Geburtshilfe, Bernburg, Germany

IPD SHARING:
Plan to Share IPD: No